CLINICAL TRIAL: NCT00005861
Title: Evaluation of Doxil as First-Line Therapy of Advanced or Recurrent Endometrial Carcinoma
Brief Title: Liposomal Doxorubicin in Treating Patients With Advanced or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067891; GOG-0086M
Record Dates: First submitted 2000-06-02; First posted 2003-05-19 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2002-08

CONDITIONS: Endometrial Cancer
Keywords: stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating women who have recurrent, stage III, or stage IV endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity and safety of doxorubicin HCl liposome in patients with advanced or recurrent endometrial cancer.
* Determine the response rate, response duration, and overall survival of these patients treated with this regimen.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 1 hour. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III, IV, or recurrent endometrial carcinoma for which curative radiotherapy or surgery is not an option
* Bidimensionally measurable disease

  * Irradiated field as only site allowed if evidence of progression since radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* LVEF normal by cardiac echocardiogram or MUGA

Other:

* No concurrent active infection
* No prior or concurrent malignancy within past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy as radiosensitizer allowed
* No prior chemotherapy for advanced or metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No prior therapy that would preclude study
* No other concurrent antineoplastic agents
* No other concurrent investigational agents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-05; Primary Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard D. Homesley, MD, Study Chair — Gynecologic Oncology Network; Paula M. Fracasso, MD, PhD — Washington University Siteman Cancer Center
Locations (10):
- United States (10):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - New England Medical Center Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Brookview Research, Inc., Nashville, Tennessee

REFERENCES:
- [Result] Homesley HD, Blessing JA, Sorosky J, Reid G, Look KY. Phase II trial of liposomal doxorubicin at 40 mg/m(2) every 4 weeks in endometrial carcinoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2005 Aug;98(2):294-8. doi: 10.1016/j.ygyno.2005.05.016. PMID 15975638